CLINICAL TRIAL: NCT02925104
Title: A Multicenter, Open Label, Phase 1 Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of INC280 Tablet Formulation With Food in Patients With cMET Dysregulated Advanced Solid Tumors.
Brief Title: A Dose Escalation Study to Assess PK, Safety and Tolerability of INC280 When Taken With Food in cMET Dysregulated Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2108; 2016-001829-14 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-02

CONDITIONS: cMET Dysegulation Advanced Solid Tumors
Keywords: cMET, INC280, food,
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INC280 (Experimental)
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280

SUMMARY:
Dose escalation study to assess PK, safety and tolerability of INC280 when taken with food in patients with cMET dysregulated advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* cMET dysregulated advanced solid tumor
* At least one measurable lesion as defined by RECIST 1.1
* Recovered from all toxicities related to prior anti-cancer therapies to grade ≤ 1
* Adequate organ function
* ECOG performance status (PS) ≤ 1

Exclusion Criteria:

* Prior treatment with crizotinib or any other cMET or HGF inhibitor
* Known hypersensitivity to any of the excipients of INC280
* Symptomatic central nervous system (CNS) metastases who are neurologically unstable
* Presence or history of a malignant disease other than the study related cancer
* Clinically significant, uncontrolled heart diseases
* Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting INC280 or patients who have not recovered from radiotherapy-related toxicities
* Major surgery within 4 weeks prior to starting INC280
* Impairment of GI function
* Patients receiving unstable or increasing doses of corticosteroids
* Patients receiving treatment with any enzyme-inducing anticonvulsant
* Pregnant or nursing (lactating) women Other protocol-related inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxiticites (DLTs) | During the first 28 days on INC280 treatment; cycle = 21 days
Frequency of DLTs | During the first 28 days on INC280 treatment
Category of DLTs | During the first 28 days on INC280 treatment
AUClast for INC280 | Treatment Cycle 1 Day 1 (C1D1), C1D7, C1D15, C2D1, C3D1
AUCtau for INC280 | C1D1, C1D7, C1D15, C2D1, C3D1
Cmax for INC280 | C1D1, C1D7, C1D15, C2D1, C3D1
Tmax | C1D1, C1D7, C1D15, C2D1, C3D1

SECONDARY OUTCOMES:
Adverse events based on CTCAE grading and other safety variables (e.g. EGC readings, physical examination, vital signs and laboratory results). | Screening, until 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Indiana University Simon Cancer Center SC, Indianapolis, Indiana, United States
- Novartis Investigative Site, Salzburg, Austria
- Novartis Investigative Site, Herlev, Denmark
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Nijmegen, Netherlands
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno V, Greil R, Yachnin J, Majem M, Wermke M, Arkenau HT, Basque JR, Nidamarthy PK, Kapoor S, Cui X, Giovannini M. Pharmacokinetics and safety of capmatinib with food in patients with MET-dysregulated advanced solid tumors. Clin Ther. 2021 Jun;43(6):1092-1111. doi: 10.1016/j.clinthera.2021.04.006. Epub 2021 May 27. PMID 34053700
- See also: Results for CINC280A2108 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17391